CLINICAL TRIAL: NCT01010009
Title: Effects of Resveratrol on Cerebral Blood Flow Parameters and Cognitive Performance in Humans: a Double-blind, Placebo-controlled, Crossover Investigation
Brief Title: The Cognitive and Cerebral Blood Flow Effects of Resveratrol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Emma Wightman, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 22P2
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Cognitive and Cerebral Blood Flow Effects of Resveratrol
Keywords: resveratrol; cerebral blood flow; NIRS; cognitive performance
MeSH Terms: interventions — Resveratrol; Silicon Dioxide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Resveratrol 250mg (Experimental)
  Interventions: Dietary Supplement: Trans- resveratrol; Other: Placebo (silica)
- Resveratrol 500mg (Experimental)
  Interventions: Dietary Supplement: Trans- resveratrol; Other: Placebo (silica)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Trans- resveratrol; Other: Placebo (silica)

INTERVENTIONS:
Dietary Supplement: Trans- resveratrol — All 24 participants who completed the study took part in 3 conditions; receiving either 250mg resveratrol, 500mg resveratrol or placebo on separate days (with a 48hr-14day wash out period between each treatment) with the order dictated by a latin square. Treatment was administered in capsule form and in a double blind manner.
  Other Names: Transmax from Biotivia.
Other: Placebo (silica) — All 24 participants who completed the study took part in 3 conditions; receiving either 250mg resveratrol, 500mg resveratrol or placebo on separate days (with a 48hr-14day wash out period between each treatment) with the order dictated by a latin square. Treatment was administered in capsule form and in a double blind manner.
  Other Names: Pharmaceutical grade silica

SUMMARY:
Research shows that resveratrol is able to induce vasodilation (and therefore blood flow) by interacting with nitric oxide (NO). Research also shows that acute administration of metabolic substrates, like oxygen and glucose, can enhance aspects of cognitive performance in young, healthy humans. The aim of this investigation was to determine if the consumption of resveratrol could modulate cerebral blood flow and if this in turn could influence cognitive performance by increasing access to blood borne metabolic fuel. Results showed that compared to placebo, after consuming 500mg pure trans-resveratrol, levels of total haemoglobin were significantly higher in the frontal cortex of young, healthy participants during cognitive task completion. Cognitive performance was not effected.

ELIGIBILITY:
Inclusion Criteria:

* Male/female,
* Healthy
* Age 18-35 years old
* Non smoker
* Proficient in English
* Not taking any herbal or prescription medications
* Not pregnant
* Does not drink more than 6 cups of coffee per day

Exclusion Criteria:

* Suffered a head injury, neurological disorder or neuro-developmental disorder
* Food allergies/intolerances

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Haskell, Study Director — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Resveratrol 250mg Then Resveratrol 500mg Then Placebo | Resveratrol 500mg Then Placebo Then Resveratrol 250mg | Placebo Then Resveratrol 250mg Then Resveratrol 500mg
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resveratrol 250mg Then Resveratrol 500mg Then Placebo | Resveratrol 500mg Then Placebo Then Resveratrol 250mg | Placebo Then Resveratrol 250mg Then Resveratrol 500mg | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 19.2 (2.2) | 21.3 (1.8) | 20 (2) | 20 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 7 | 20
  Male | 2 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Modulation of Levels of Total Haemoglobin
Description: This outcome measure provides the change from baseline values (in µmol/L) of total levels of haemoglobin during the 46-81 min post dose testing period. This was measured in the frontal cortex by near infrared spectroscopy (NIRS).
Time Frame: 0-81 mins (absorption period=1- 45 mins , post dose period 46- 81 mins)
Population: NIRS data was analysed for all participants who completed the trial and who were not noted as having significantly high or low readings during data collection.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Resveratrol 250mg | Resveratrol 500mg | Placebo
Number analyzed (Participants) | 22 | 22 | 22
µmol/L | 1.9 (0.9) | 2.4 (0.8) | 1.2 (0.1)
Statistical Analysis 1: Comparison: Resveratrol 250mg vs Placebo; Data was analysed by omnibus ANOVA with a priori planned comparisons utilizing the mean squares error term from this ANOVA; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Resveratrol 500mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: Number of Participants With Significant Modulation of Cognitive Performance
Description: This outcome measure assessed any significant modulation of cognitive task performance during the 46-81 min post dose period. The cognitive tasks utilized were cognitively demanding computer based, numerical tasks which assessed working memory. Significant modulation is defined as significant difference between baseline and post-dose task performance.
Time Frame: 46-81 mins post dose
Population: Cognitive performance data was analysed for all subjects who completed the trial. If data was not utilized in the final analysis then this was either due to technical issues (i.e. the computer did not save data) or it was clear that the participant had not engaged with the task/s.
Measure: Number; unit: Participants
Arm/Group | Resveratrol 250mg | Resveratrol 500mg | Placebo
Number analyzed (Participants) | 22 | 22 | 22
Participants | 0 (0) | 0 (0) | 0 (0)
Statistical Analysis 1: Comparison: Resveratrol 250mg vs Placebo; Performance on each cognitive task was assessed via omnibus ANOVA with a priori planned comparisons; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Resveratrol 500mg vs Placebo; Performance on each cognitive task was assessed via omnibus ANOVA with a priori planned comparisons; Test type: Superiority or Other; p > 0.05, ANOVA

3. Primary Outcome: Modulation of Deoxygenated Levels of Haemoglobin
Description: This outcome measure provides the change from baseline values (in µmol/L) of levels of deoxygenated haemoglobin during the 46-81 min post dose testing period. This was measured in the frontal cortex by near infrared spectroscopy (NIRS).
Time Frame: 0-81 mins (absorption period=1- 45 mins , post dose period 46- 81 mins)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Resveratrol 250mg | Resveratrol 500mg | Placebo
Number analyzed (Participants) | 22 | 22 | 22
µmol/L | 0.4 (0.2) | 0.2 (0.11) | -0.2 (0.1)
Statistical Analysis 1: Comparison: Resveratrol 250mg vs Placebo; An omnibus ANOVA was carried out with a priori planned comparisons using the mean squares error term from this ANOVA; Test type: Superiority or Other; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: Resveratrol 500mg vs Placebo; An omnibus ANOVA was carried out with a priori planned comparisons using the mean squares error term from this ANOVA; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | Resveratrol 250mg | Resveratrol 500mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes